CLINICAL TRIAL: NCT03223467
Title: Effect of Bariatric Surgery on Obstructive Sleep Apnea and Predictors for the Severity of Obstructive Sleep Apnea
Brief Title: Obstructive Sleep Apnea, Predictors and Bariatric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Geltrude Mingrone, Professor, Catholic University of the Sacred Heart
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OSA2012
Record Dates: First submitted 2017-07-14; First posted 2017-07-21 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Obesity; Obstructive Sleep Apnea; Bariatric Surgery Candidate
Keywords: Obesity; Obstructive sleep apnea; Bariatric surgery candidate; Metabolic syndrome
MeSH Terms: conditions — Obesity; Sleep Apnea, Obstructive; Metabolic Syndrome | interventions — Bariatric Surgery

STUDY DESIGN:
Intervention Model Description: Patients in this study underwent either gastric bypass, gastric sleeve or biliopancreatic diversion. Some patient choose not to undergo bariatric surgery and function as a control arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Biliopancreatic diversion (Active Comparator): Study participants will undergo biliopancreatic diversion which is a type of bariatric surgery where a part of the stomach are removed and the remaining stomach is attached to a distal segment of the small intestine.
  Interventions: Procedure: Bariatric surgery
- Gastric sleeve (Active Comparator): Study participants will undergo sleeve gastrectomy which is a restrictive form av bariatric surgery where the size of the stomach is reduced.
  Interventions: Procedure: Bariatric surgery
- Gastric bypass (Active Comparator): Study participants will undergo gastric bypass which is a type of bariatric surgery where a small pouch of the stomach is created and attached to a segment of the small intestine.
  Interventions: Procedure: Bariatric surgery
- No intervention (No Intervention): Study participants that do not want to undergo surgical treatment.

INTERVENTIONS:
Procedure: Bariatric surgery — Bariatric surgery includes several different types of surgical procedures used to achieve weight loss.
  Arms: Biliopancreatic diversion; Gastric bypass; Gastric sleeve

SUMMARY:
Obstructive sleep apnea is defined as a repetitive collapse of the pharynx during sleep (Malhotra, et al. 2012) which cases intermittent hypoxia. Snoring, witnessed apnea, fatigue and morning headache are symptoms of the disease which has severe health effect (Malhotra. et al. 2012) including increased mortality risk (Ensrud. et al. 2012) and effects on quality of life (Kuhn. et al. 2017).

Obesity, male sex and age are all risk factors for obstructive sleep apnea (Schwartz. et al. 2010, Edwards. et al. 2010) . Bariatric surgery is known to be a good treatment to achieve a sustained weight loss but the long term effects of bariatric treatment of obstructive sleep apnea is not well studied. The aim of this study is therefore to study the long effects of bariatric surgery as a treatment for obstructive sleep apnea and to find predictors that can be used to predict the severity of the disease.

DETAILED DESCRIPTION:
Obstructive sleep apnea is defined as a repetitive collapse of the pharynx during sleep (Malhotra, et al. 2012) which cases intermittent hypoxia. Snoring, witnessed apnea, fatigue and morning headache are symptoms of the disease which has severe health effect (Malhotra. et al. 2012) including increased mortality (Ensrud. et al. 2012) and effects on quality of life (Kuhn. et al. 2017). Hence, identifying and treat obstructive sleep apnea are important.

Obesity, male sex and age are all risk factors for obstructive sleep apnea (Schwartz et. al. 2010, Edwards. et. al. 2010) . Bariatric surgery is known to be a good treatment to achieve a sustained weight loss but the long term effects of bariatric treatment of obstructive sleep apnea is not well studied. The aim of this study is therefore to study the long effects of bariatric surgery as a treatment for obstructive sleep apnea and to find predictors that can be used to predict the severity of the disease.

Eighty-six patients with obesity have been recruited at the Catholic University hospital in Rome, Italy during 2012 when patients were enrolled during their evaluation for bariatric surgery. At baseline, the patient underwent fasting blood chemistry, anthropometric measurements and overnight polysomnography. The patients also underwent a 3 hour oral glucose tolerance test in order to determinate glucose tolerance (normal glucose tolerance, impaired glucose tolerance and type 2 diabetes mellitus). Patient then received treatment with bariatric surgery (gastric sleeve, biliopancreatic diversion or gastric bypass) during 2012-2013 or decided not to undergo bariatric surgery.

Patient will undergo follow-up during 2016-2017 where fasting blood chemistry, anthropometric measurements and overnight polysomnography will be assessed. The patient will also undergo a 3 hour oral glucose tolerance test.

The effects of bariatric surgery on obstructive sleep apnea will then be evaluated. Differences in the treatment effect between the different bariatric surgical procedures will be studied. Patients characteristics at baseline, such as weight, height, BMI and components of the metabolic syndrome and their association to the severity of obstructive sleep apnea will be studied in order to find predictors for the severity of the disease.

ELIGIBILITY:
Inclusion Criteria:

* BMI above 30 kg/m2
* Age between 20 and 70 years
* Willingness to understand the protocol and willingness to participate in the study

Exclusion Criteria:

* Exclusion criteria is severe co-morbidities that would prevent the patients to undergo bariatric surgery. Such as severe anemia, severe heart failure, active or previous malignancies the last 5 years. Myocardial infarction or unstable angina pectoris the last 6 months. Pregnancy. Suspected poor compliance. Drug or alcohol abuse. Major gastrointestinal disease.
* Inability to undergo polysomnography.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2012-01-04 (Actual); Primary Completion 2017-12-30 (Actual); Study Completion 2017-12-30 (Actual)

PRIMARY OUTCOMES:
Change in severity of obstructive sleep apnea measured by a overnight cardio-respiratory monitoring before and 5 years after bariatric surgery. | 5 years
  The effect of bariatric surgery as a treatment of obstructive sleep apnea in patients with obesity will be evaluated as the change in obstructive sleep apnea severity. To address this aim a overnight cardio-respiratory monitoring with a Vital Night 8 device (Vital Aire, Milan, Italy) will be performed before and 5 years after bariatric surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Geltrude Mingrone, MD. PhD., Principal Investigator — The Catholic University of the Sacred Heart

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Malhotra A, White DP. Obstructive sleep apnoea. Lancet. 2002 Jul 20;360(9328):237-45. doi: 10.1016/S0140-6736(02)09464-3. PMID 12133673
- [Background] Ensrud KE, Blackwell TL, Ancoli-Israel S, Redline S, Cawthon PM, Paudel ML, Dam TT, Stone KL. Sleep disturbances and risk of frailty and mortality in older men. Sleep Med. 2012 Dec;13(10):1217-25. doi: 10.1016/j.sleep.2012.04.010. Epub 2012 Jun 15. PMID 22705247
- [Background] Kuhn E, Schwarz EI, Bratton DJ, Rossi VA, Kohler M. Effects of CPAP and Mandibular Advancement Devices on Health-Related Quality of Life in OSA: A Systematic Review and Meta-analysis. Chest. 2017 Apr;151(4):786-794. doi: 10.1016/j.chest.2017.01.020. Epub 2017 Jan 24. PMID 28130044
- [Background] Schwartz AR, Patil SP, Squier S, Schneider H, Kirkness JP, Smith PL. Obesity and upper airway control during sleep. J Appl Physiol (1985). 2010 Feb;108(2):430-5. doi: 10.1152/japplphysiol.00919.2009. Epub 2009 Oct 29. PMID 19875707
- [Background] Edwards BA, O'Driscoll DM, Ali A, Jordan AS, Trinder J, Malhotra A. Aging and sleep: physiology and pathophysiology. Semin Respir Crit Care Med. 2010 Oct;31(5):618-33. doi: 10.1055/s-0030-1265902. Epub 2010 Oct 12. PMID 20941662